CLINICAL TRIAL: NCT03537274
Title: Comparison of Polyethylene Glycol-Interferon Alfa-2B (PEG-Intron, SCH 54031) vs. Interferon Alfa-2B for Treatment of Adult Subjects With Chronic Hepatitis C Not Previously Treated With Interferon: Dose Finding Study
Brief Title: Efficacy of Polyethylene Glycol-Interferon Alfa-2B (PEG-Intron, SCH 54031) Compared to Interferon Alfa-2B in Participants With Chronic Hepatitis C (MK-4031-016)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C97010; MK-4031-016 (Other: Merck Protocol Number); C97010 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Interferon alpha-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PEG-Intron, 0.5 mg/kg (Experimental): PEG-Intron administered once weekly (QW) for 48 weeks at 0.5 mg/kg by subcutaneous (SC) injection.
  Interventions: Biological: PEG-Intron
- PEG-Intron, 1.0 mg/kg (Experimental): PEG-Intron administered QW for 48 weeks at 1.0 mg/kg by SC injection.
  Interventions: Biological: PEG-Intron
- PEG-Intron, 1.5 mg/kg (Experimental): PEG-Intron administered QW for 48 weeks at 1.5 mg/kg by SC injection.
  Interventions: Biological: PEG-Intron
- Interferon Alfa-2b (Active Comparator): Interferon Alfa-2b administered three times per week (TIW) for 48 weeks at 3 million international units (MIU) by SC injection.
  Interventions: Biological: Interferon Alfa-2B

INTERVENTIONS:
Biological: PEG-Intron — PEG-Intron is administered QW for 48 weeks by SC injection at 0.5, 1.0, and 1.5 mg/kg body weight. Body weight obtained at the baseline visit is used to calculate dosing.
  Other Names: SCH 54031
  Arms: PEG-Intron, 0.5 mg/kg; PEG-Intron, 1.0 mg/kg; PEG-Intron, 1.5 mg/kg
Biological: Interferon Alfa-2B — Interferon alfa-2b is administered TIW for 48 weeks by SC injection at 3 MIU regardless of participant body weight.
  Arms: Interferon Alfa-2b

SUMMARY:
This study will determine the efficacy of PEG-Intron (SCH 54031) in participants with chronic Hepatitis C virus (HCV) infection who have not been previously treated with interferon. Participants are randomized to receive one of three doses of PEG-Intron (0.5, 1.0, and 1.5 mg/kg) or Interferon Alfa-2B for 48 weeks. The primary objective of this study is to evaluate the efficacy of PEG-Intron (compared to Interferon Alfa-2B) with respect to response based on loss of detectable HCV ribonucleic acid (HCV-RNA) and normalization of alanine transaminase (ALT) level after 24 weeks of therapy and at 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Be serum positive for hepatitis C virus.
* Have liver biopsy within 1 year prior to entry, with a pathology report confirming a histological diagnosis consistent with chronic hepatitis.
* Have one abnormal historic ALT at least 6 months prior to screening, with elevated ALT at entry.
* Have compensated liver disease, testing negative for HIV and serum hepatitis B surface antigen (HBsAg) at entry.
* If male or female of childbearing potential, be practicing adequate contraception during treatment.

Exclusion Criteria:

* Be female who is currently pregnant or nursing.
* Have prior treatment with any interferon.
* Have suspected hypersensitivity to alpha interferon.
* Have participated in any other clinical trial within 30 days of entry
* Have received treatment with any investigational drug within 30 days of entry.
* Have received prior treatment for hepatitis with any other antiviral or immunomodulatory drug within the previous 2 years.
* Have any other cause for the liver disease other than chronic hepatitis C including but not limited to: co-infection with hepatitis B virus; Hemochromatosis; alpha-1 antitrypsin deficiency; Wilson's disease; autoimmune hepatitis; alcoholic liver disease; obesity-induced liver disease; and drug-related liver disease.
* Have hemophilia or any other condition that would prevent the participant from having a liver biopsy, including anticoagulant therapy.
* Have hemoglobinopathies (e.g., Thalassemia)
* Have evidence of advanced liver disease such as history or presence of ascites, bleeding varices, spontaneous encephalopathy.
* Have received organ transplants.
* Have a preexisting psychiatric condition, especially severe depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or attempt.
* Have central nervous system trauma or active seizure disorders requiring medication.
* Have significant cardiovascular dysfunction within the past 6 months (e.g., angina, congestive heart failure, recent myocardial infarction, severe hypertension or significant arrhythmia).
* Have poorly controlled diabetes mellitus.
* Have chronic pulmonary disease (e.g., chronic obstructive pulmonary disease).
* Have immunologically mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], rheumatoid arthritis, idiopathic thrombocytopenia purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical cryoglobulinemia with vasculitis).
* Have any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids.
* Have history of substance abuse, such as alcohol, intravenous drugs and inhaled drugs.
* Have clinically significant retinal abnormalities.
* Be unable to abstain from the consumption of alcohol.
* Have any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Actual)
Dates: Start 1997-08-05 (Actual); Primary Completion 1999-07-23 (Actual); Study Completion 1999-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 1224 participants with chronic Hepatitis C virus (HCV) infection were randomized, with 1219 receiving study treatment.
Period: Overall Study
Arm/Group | PEG-Intron, 0.5 mg/kg | PEG-Intron, 1.0 mg/kg | PEG-Intron, 1.5 mg/kg | Interferon Alfa-2b
Started | 315 | 298 | 304 | 307
Treated | 315 | 297 | 304 | 303
Completed | 255 | 229 | 228 | 231
Not Completed | 60 | 69 | 76 | 76

BASELINE CHARACTERISTICS:
Population: Includes all randomized participants receiving ≥1 dose of study treatment.
Groups:
- PEG-Intron, 0.5 mg/kg: PEG-Intron administered QW for 48 weeks at 0.5 mg/kg by SC injection.
- Interferon Alfa-2b: Interferon Alfa-2b administered TIW for 48 weeks at 3 MIU by SC injection.
- Total: Total of all reporting groups
Arm/Group | PEG-Intron, 0.5 mg/kg | PEG-Intron, 1.0 mg/kg | PEG-Intron, 1.5 mg/kg | Interferon Alfa-2b | Total
Number analyzed (Participants) | 315 | 297 | 304 | 303 | 1219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (9.4) | 43.7 (9.5) | 42.9 (8.7) | 42.6 (9.2) | 43.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 109 | 114 | 96 | 449
  Male | 185 | 188 | 190 | 207 | 770

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Responder Status at 24 Weeks of Treatment
Description: The number of participants achieving responder status at 24 weeks of treatment was assessed. A participant was classified as a responder if, at 24 weeks of treatment, they met both of the following criteria: 1) HCV-Ribonucleic Acid (RNA) negative (defined as <100 copies/mL serum by quantitative polymerase chain reaction [qPCR] assay); and 2) alanine transaminase (ALT) level normal.
Time Frame: Up to 24 weeks
Population: Includes all randomized participants receiving ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PEG-Intron, 0.5 mg/kg | PEG-Intron, 1.0 mg/kg | PEG-Intron, 1.5 mg/kg | Interferon Alfa-2b
Number analyzed (Participants) | 315 | 297 | 304 | 303
Participants | 80 | 87 | 90 | 59
Statistical Analysis 1: Comparison: PEG-Intron, 0.5 mg/kg vs Interferon Alfa-2b; Test type: Superiority; p = 0.078, Chi-squared
Statistical Analysis 2: Comparison: PEG-Intron, 1.0 mg/kg vs Interferon Alfa-2b; Test type: Superiority; p = 0.005, Chi-squared
Statistical Analysis 3: Comparison: PEG-Intron, 1.5 mg/kg vs Interferon Alfa-2b; Test type: Superiority; p = 0.004, Chi-squared

2. Primary Outcome: Number of Participants Achieving Sustained Responder Status at 24 Weeks of Follow-up
Description: The number of participants achieving sustained responder status at 24 weeks of follow-up was assessed. A participant was classified as a sustained responder if, at 24 weeks of follow-up, they met both of the following criteria: 1) HCV-RNA negative (defined as <100 copies/mL serum by qPCR assay); and 2) ALT level normal.
Time Frame: Up to 72 weeks (up to 48 weeks treatment and 24 weeks follow-up)
Population: Includes all randomized participants receiving ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PEG-Intron, 0.5 mg/kg | PEG-Intron, 1.0 mg/kg | PEG-Intron, 1.5 mg/kg | Interferon Alfa-2b
Number analyzed (Participants) | 315 | 297 | 304 | 303
Participants | 52 | 70 | 69 | 37
Statistical Analysis 1: Comparison: PEG-Intron, 0.5 mg/kg vs Interferon Alfa-2b; Test type: Superiority; p = 0.128, Chi-squared
Statistical Analysis 2: Comparison: PEG-Intron, 1.0 mg/kg vs Interferon Alfa-2b; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: PEG-Intron, 1.5 mg/kg vs Interferon Alfa-2b; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 72 weeks (up to 48 weeks treatment and 24 weeks of follow-up)
Description: Analysis population includes all randomized participants receiving ≥1 dose of study treatment.
Groups:
- PEG-Intron, 0.5 mg/kg: PEG-Intron administered QW for 48 weeks at 0.5 mg/kg SC injection.
Arm/Group | PEG-Intron, 0.5 mg/kg | PEG-Intron, 1.0 mg/kg | PEG-Intron, 1.5 mg/kg | Interferon Alfa-2b
All-Cause Mortality (participants affected / at risk) | 1/315 | 0/297 | 0/304 | 2/303
Serious Adverse Events (participants affected / at risk) | 37/315 | 32/297 | 31/304 | 29/303
Other Adverse Events (participants affected / at risk) | 306/315 | 291/297 | 296/304 | 293/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron, 0.5 mg/kg (N=315) | PEG-Intron, 1.0 mg/kg (N=297) | PEG-Intron, 1.5 mg/kg (N=304) | Interferon Alfa-2b (N=303)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic vein thrombosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal exudates (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Douglas' abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body fat disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron, 0.5 mg/kg (N=315) | PEG-Intron, 1.0 mg/kg (N=297) | PEG-Intron, 1.5 mg/kg (N=304) | Interferon Alfa-2b (N=303)
Neutropenia (Blood and lymphatic system disorders) | 13 (26) | 18 (37) | 25 (36) | 7 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (13) | 19 (37) | 15 (17) | 1 (1)
Hypothyroidism (Endocrine disorders) | 10 (12) | 18 (22) | 15 (19) | 11 (13)
Abdominal discomfort (Gastrointestinal disorders) | 12 (16) | 17 (20) | 15 (18) | 15 (18)
Abdominal pain (Gastrointestinal disorders) | 28 (37) | 24 (31) | 19 (20) | 14 (16)
Abdominal pain upper (Gastrointestinal disorders) | 48 (75) | 38 (51) | 37 (54) | 33 (39)
Diarrhoea (Gastrointestinal disorders) | 53 (75) | 58 (90) | 69 (103) | 50 (70)
Dry mouth (Gastrointestinal disorders) | 11 (12) | 12 (13) | 25 (28) | 12 (13)
Dyspepsia (Gastrointestinal disorders) | 16 (20) | 11 (13) | 12 (20) | 15 (17)
Nausea (Gastrointestinal disorders) | 73 (114) | 83 (128) | 83 (130) | 64 (95)
Vomiting (Gastrointestinal disorders) | 22 (29) | 23 (36) | 23 (33) | 20 (22)
Asthenia (General disorders) | 42 (89) | 40 (89) | 50 (120) | 41 (63)
Chest pain (General disorders) | 12 (14) | 17 (20) | 7 (10) | 8 (8)
Chills (General disorders) | 106 (140) | 120 (162) | 133 (184) | 99 (125)
Fatigue (General disorders) | 160 (279) | 164 (283) | 159 (287) | 170 (295)
Influenza like illness (General disorders) | 57 (74) | 66 (95) | 76 (113) | 59 (78)
Injection site erythema (General disorders) | 135 (189) | 120 (166) | 122 (164) | 47 (49)
Malaise (General disorders) | 20 (41) | 27 (43) | 24 (86) | 21 (28)
Pain (General disorders) | 55 (89) | 61 (87) | 60 (90) | 50 (64)
Pyrexia (General disorders) | 96 (141) | 124 (191) | 127 (206) | 86 (106)
Hepatomegaly (Hepatobiliary disorders) | 20 (22) | 16 (17) | 16 (18) | 10 (12)
Liver tenderness (Hepatobiliary disorders) | 12 (12) | 10 (12) | 16 (17) | 9 (10)
Bronchitis (Infections and infestations) | 15 (24) | 18 (19) | 13 (19) | 10 (12)
Influenza (Infections and infestations) | 17 (21) | 19 (22) | 20 (23) | 22 (29)
Nasopharyngitis (Infections and infestations) | 36 (45) | 21 (31) | 27 (33) | 24 (30)
Sinusitis (Infections and infestations) | 26 (33) | 21 (22) | 27 (37) | 19 (29)
Upper respiratory tract infection (Infections and infestations) | 20 (23) | 12 (14) | 9 (10) | 14 (22)
Weight decreased (Investigations) | 34 (45) | 36 (45) | 74 (91) | 42 (46)
Decreased appetite (Metabolism and nutrition disorders) | 33 (39) | 59 (72) | 76 (86) | 49 (60)
Arthralgia (Musculoskeletal and connective tissue disorders) | 78 (145) | 71 (116) | 86 (159) | 73 (124)
Back pain (Musculoskeletal and connective tissue disorders) | 46 (58) | 57 (81) | 48 (78) | 56 (89)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 (34) | 15 (21) | 11 (15) | 12 (21)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (14) | 17 (24) | 8 (10) | 12 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 111 (212) | 107 (178) | 135 (249) | 114 (187)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (31) | 31 (45) | 22 (34) | 20 (22)
Disturbance in attention (Nervous system disorders) | 20 (27) | 22 (29) | 21 (23) | 16 (19)
Dizziness (Nervous system disorders) | 29 (34) | 38 (43) | 45 (58) | 34 (51)
Headache (Nervous system disorders) | 192 (445) | 200 (481) | 195 (492) | 177 (351)
Anxiety (Psychiatric disorders) | 32 (59) | 30 (51) | 25 (34) | 33 (53)
Depression (Psychiatric disorders) | 73 (135) | 72 (114) | 74 (116) | 66 (112)
Insomnia (Psychiatric disorders) | 51 (73) | 74 (101) | 58 (82) | 64 (105)
Irritability (Psychiatric disorders) | 65 (92) | 53 (76) | 57 (84) | 74 (106)
Libido decreased (Psychiatric disorders) | 9 (9) | 6 (7) | 10 (13) | 17 (19)
Nervousness (Psychiatric disorders) | 14 (20) | 15 (22) | 10 (15) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (28) | 25 (27) | 30 (36) | 16 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (25) | 12 (14) | 15 (15) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 17 (20) | 16 (18) | 16 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 64 (75) | 68 (82) | 104 (113) | 67 (78)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (23) | 33 (38) | 29 (33) | 27 (30)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 16 (21) | 13 (14) | 17 (23) | 13 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 30 (38) | 37 (45) | 28 (30) | 22 (28)
Rash (Skin and subcutaneous tissue disorders) | 22 (27) | 21 (24) | 24 (27) | 18 (19)
Hot flush (Vascular disorders) | 8 (9) | 16 (17) | 7 (8) | 6 (7)

LIMITATIONS AND CAVEATS:
Adverse Event (AE) Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 21.0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide the Sponsor thirty (30) days prior to submission for publication or presentation, copies of abstracts or manuscripts for publication which report project results. The Sponsor shall have editorial rights with respect to Publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to (a) proprietary information and, (b) the accuracy of the information contained in the Publication.